CLINICAL TRIAL: NCT05533190
Title: Real World Testing of an Artificial Intelligence-enabled App as an Early Intervention and Support Tool in the Mental Health Referral Care Pathway
Brief Title: Clinical Investigation of Wysa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); Imperial College London (Other); University of Warwick (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Associate Professor of eHealth, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM1000411
Record Dates: First submitted 2022-09-01; First posted 2022-09-08 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Issue; Anxiety; Depressive Symptoms
Keywords: Artificial Intelligence; Mental Health; Telemedicine; Conversational Agent
MeSH Terms: conditions — Anxiety Disorders; Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to the intervention condition or a standard care waitlist control condition.
Masking Description: Due to the nature of the intervention, no blinding of participants will be possible in the study, as all participants will know whether or not they are using the app. Clinical treatment teams will also not be blinded as they will know through the electronic patient record if a participant has received the intervention. The evaluation team will be blinded to treatment using the randomisation algorithm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wysa AI chatbot mental health app (Experimental): Wysa is a guided self-help and triaging tool delivered to patients via an app or widget. It uses Natural Language Processing to understand individuals' written inputs but not to generate responses. Wysa makes use of a wide range of clinically underpinned modules whilst gamification, clinical outcome measures and AI promotes engagement, improving efficacy and triage and reducing the cost of scale.
  Interventions: Device: Wysa AI chatbot mental health app
- Waitlist control (No Intervention): The intervention will be compared against a waitlist group. This comparator was selected to compare Wysa to the current standard of care for patients waiting for standard IAPT assessment and treatment.

INTERVENTIONS:
Device: Wysa AI chatbot mental health app — Wysa is a guided self-help and triaging tool delivered to patients via an app. It includes a chatbot and makes use of a wide range of clinically underpinned modules to provide mental health support.
  Arms: Wysa AI chatbot mental health app

SUMMARY:
Mental health concerns are a large burden for individuals, healthcare systems, and the economy. Over a million people are referred to UK mental health services each year, but more than half only receive one session of workbook-based support. Many others have to wait over 12 weeks for assessment and treatment. Wysa is a digital health app with over 3 million users that uses an artificial intelligence (AI) chatbot and a series of self-care exercises to provide mental health support and to help people develop strategies to manage their mental health and improve their resilience.

This project aims to examine the impact of using Wysa on patients' symptoms of anxiety and depression during the referral process for standard UK mental health services. Patients will be given access to Wysa at the point of referral to the Improving Access to Psychological Therapies (IAPT) programme and can begin to explore the self-support tools, while they are on the waitlist for assessment and treatment. The investigators will gather a group of patients and members of the public to contribute to the recruitment of patients for the study, the methods we use to evaluate Wysa, and to provide insights on how best to share the results of our study with the general public.

The investigators will use the standard IAPT measures of anxiety and depression to look at the effect of using Wysa patients' mental well-being. These questionnaires will be provided through the app and the results will be compared with a waitlist control group. The investigators will examine whether Wysa can identify people who are experiencing severe mental health difficulties so that they can be provided with additional support. Users' levels of engagement with Wysa will be assessed and some participants will be randomly selected to do an interview so the investigators can get a better understanding of what people liked and disliked about using the app and why. Finally, the investigators will be evaluating the cost-effectiveness of Wysa compared with usual care.

The investigators expect that the study will show that Wysa helps reduce symptoms of anxiety and depression in people who are on the waiting list for IAPT. If the study shows this positive impact, this will provide evidence to support the use of Wysa to improve the accessibility of mental health support in clinical pathways. The investigators will be publishing the results of our study in academic journals as well as in more generally accessible platforms.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Aged 18 years or older;
* Ability to speak English to a secondary school standard;
* Own a mobile device capable of supporting Wysa;
* A valid email address;
* Referred or self-referred to proceed through the standard IAPT care pathway.

Exclusion Criteria:

* Patients ineligible for the standard IAPT care pathway;
* Patients with previous and current known major mental illness such as Schizophrenia, severe depression, any co-morbid neurological or neuro-psychiatric condition such as epilepsy;
* Patients with current psychosis or a history of psychotic symptoms within the last 6 months;
* Patients with suicidal ideation;
* Patients scoring > 15 points on PHQ 9;
* Patients scoring > 15 points on GAD-7;
* Patients with significant cognitive disorders;
* Patients with noted neurodevelopmental conditions such as autism or ADHD;
* Patients previously diagnosed with a personality disorder;
* Patients who been under the care of CMHT or a specialised mental health services in the last 2 years;
* Patients who failed IAPT previously;
* Patients with referrals for specialist presentations of pre-existing, diagnosed conditions requiring a specialised assessment beyond the standard clinical pathway;
* Incapable of self-consent;
* In a dependent/unequal relationship with the research or care teams or any PPI representatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-07-23 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Shankar, FRCPsych, Principal Investigator — University of Plymouth
Locations (2):
- United Kingdom (2):
  - University of Plymouth, Plymouth, Devon
  - Central North West London NHS, London

IPD SHARING:
Plan to Share IPD: No
Only the Academic CIs and their research staff will have access to research data.

REFERENCES:
- [Derived] Milne-Ives M, Homer SR, Andrade J, Meinert E. Mapping the Process of Engagement With Digital Health Interventions: A Cross-Case Synthesis. Mayo Clin Proc Innov Qual Outcomes. 2025 May 27;9(3):100625. doi: 10.1016/j.mayocpiqo.2025.100625. eCollection 2025 Jun. PMID 40503087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Started | 53 | 23
Completed | 30 | 16
Not Completed | 23 | 7
Not completed — Lost to Follow-up | 19 | 7
Not completed — Failed to download app | 1 | 0
Not completed — Thought app was a scam | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control | Total
Number analyzed (Participants) | 30 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (14.4) | 37.1 (15.8) | 36.3 (14.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 11 | 29
  Male | 10 | 4 | 14
  Transgender female | 1 | 1 | 2
  Declined to respond | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Asian British | 3 | 1 | 4
  Not known | 1 | 2 | 3
  Other ethnic groups | 4 | 5 | 9
  White | 21 | 8 | 29
  Black or Black British | 1 | 0 | 1
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Score on the PHQ-9, total scores range from 0 to 27 (higher scores indicated more severe depression)
  units on a scale | 11.9 (5.07) | 11.0 (4.38) | 11.6 (4.81)
GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Score on the GAD-7, total scores range from 0 to 21 (higher scores indicated more severe anxiety)
  units on a scale | 11.3 (4.92) | 11.9 (4.92) | 11.5 (4.87)

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Score on the PHQ-9, total scores range from 0 to 27 (higher scores indicated more severe depression)
Time Frame: 3 months post-randomisation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Number analyzed (Participants) | 30 | 16
units on a scale | 9.28 (6.56) | 8.41 (3.82)

2. Secondary Outcome: Anxiety Severity
Description: Score on the GAD-7, total scores range from 0 to 21 (higher scores indicated more severe anxiety)
Time Frame: 3 months post-randomisation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Number analyzed (Participants) | 30 | 16
units on a scale | 8.98 (6.13) | 8.19 (3.22)

3. Secondary Outcome: Crisis Identification
Description: Planned to compare number of users identified by the app for escalation of care compared to the number of patients in the control group who access A&E or out-of-hours services while waiting for treatment; this was not possible, data reported reflect risk events triggered by Wysa or the participant in-app
Time Frame: 3 months post-randomisation
Population: Waitlist control group was not analysed for "Users triggered in-app escalation" or "App identified and flagged suicidal language" because these participants did not have access to the app
Measure: Number; unit: participants
Groups:
- Waitlist Control: Participants following standard care pathway
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Number analyzed (Participants) | 30 | 16
participants
  Users triggered in-app escalation: number analyzed (Participants) | 30 | 0
  Users triggered in-app escalation | 4 |
  App identified and flagged suicidal language: number analyzed (Participants) | 30 | 0
  App identified and flagged suicidal language | 1 |
  Self-reports to the service or crisis service reports (iaptus record) | 0 | 0

4. Secondary Outcome: Uptake Rates
Description: Uptake rates of participants randomised into intervention group
Time Frame: 3 months post-randomisation
Population: Participants randomly assigned to intervention group
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Standard care pathway
Arm/Group | Wysa AI Chatbot Mental Health App | Control Group
Number analyzed (Participants) | 53 | 23
Participants | 30 | 16

5. Secondary Outcome: Dropout Rates
Description: Dropout rates of participants who are randomised into intervention group and start using the app
Time Frame: 3 months post-randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Number analyzed (Participants) | 53 | 23
Participants | 23 | 7

6. Secondary Outcome: Use of the App
Description: Participant engagement with the app (whether it was used at all based on app usage data)
Time Frame: 3-7 months post-randomisation
Population: Participants assigned to Wysa group
Measure: Count of Participants; unit: Participants
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 30
Participants
  Engaged with Wysa | 18
  Did not engage with Wysa | 12

7. Secondary Outcome: Engagement
Description: Qualitative feedback from semi-structured interviews about engagement with the app
Time Frame: 3-7 months post randomisation
Population: Participants in the Wysa group who completed semi-structured interviews - the numbers reported are counts of the number of participants who expressed a particular theme generated from the thematic analysis
Measure: Number; unit: participants
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 4
participants
  Minimal transfer of skills beyond app | 4
  Reminders helped prompt use but app was easy to ignore | 4
  Varying patterns of use for individuals | 4
  Decrease in use over time | 2

8. Secondary Outcome: Patient Perceptions of Acceptability
Description: Qualitative feedback from semi-structured interviews about the acceptability of the app
Time Frame: 3-7 months post randomisation
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 4
participants
  App did not meet all needs; not long-term solution or replacement for therapy | 4
  Easy to use but a bit overwhelming | 4
  Limited chatbot frustrated users | 4
  Range of resources were useful for users | 4
  Suggestions for improvement | 3
  Tone affected user connection with app | 3
  Tool was exciting and a relief because of accessible support and expected benefit | 4
  Trustworthiness shaped by source credibility and personal experience | 4

9. Secondary Outcome: General Health State
Description: 5-level EQ-5D version (EQ-5D-5L) which measures health-related quality of life via 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual scale - total survey scores were calculated and can range from 5 to 125 (higher scores indicate more severe health problems). A single index was obtained by transforming the ordinal survey responses using the 'eq5d' package in R.
  Range: The EQ-5D index score typically ranges from -0.594 to 1 (depending on the country-specific value set used).
  Interpretation:
  1.000 represents full health (the best possible outcome). 0.000 represents a health state equivalent to death (neutral point). Negative values (e.g., -0.594) indicate health states perceived as worse than death.
  Higher index values indicate better health outcomes, while lower values represent poorer health states.
  https://euroqol.org/wp-content/uploads/2023/11/EQ-5D-5LUserguide-23-07.pdf
Time Frame: Measured at baseline and 3 months post-randomisation
Population: Not all participants completed the follow-up assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
Number analyzed (Participants) | 30 | 16
units on a scale
  Baseline | 0.681 (0.163) | 0.607 (0.235)
  12 weeks: number analyzed (Participants) | 21 | 13
  12 weeks | 0.688 (0.174) | 0.644 (0.192)

10. Secondary Outcome: Type of App Usage - Exercises Completed
Description: Frequency and duration of app use
Time Frame: 3 months post-randomisation
Population: Participants assigned to Wysa intervention group; data from some participants was missing if they did not use that feature.
Measure: Mean (Standard Deviation); unit: Exercises completed
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 30
Exercises completed | 7.11 (7.79)

11. Secondary Outcome: Type of App Usage - Sessions Completed
Description: Frequency and duration of app use
Time Frame: 3 months post-randomisation
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Sessions completed
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 18
Sessions completed | 24.3 (29.8)

12. Secondary Outcome: Type of App Usage - Messages to Chatbot
Description: Frequency and duration of app use
Time Frame: 3 months post-randomisation
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Messages to chatbot
Arm/Group | Wysa AI Chatbot Mental Health App
Number analyzed (Participants) | 18
Messages to chatbot | 227 (319)

ADVERSE EVENTS:
Time Frame: 3 months post-randomisation
Description: We have included risk events for the purpose of clarity; appropriate signposting was provided for all of the users with risk events.
Arm/Group | Wysa AI Chatbot Mental Health App | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/16
Other Adverse Events (participants affected / at risk) | 5/30 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Wysa AI Chatbot Mental Health App (N=30) | Waitlist Control (N=16)
Suicidal language (General disorders) | 1 | 0 — Suicidal language used by participants in their discussions with the chatbot was detected by the app and flagged
User-triggered escalation in app (General disorders) | 4 | 0 — User escalation within the app was captured as a risk event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05533190/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05533190/SAP_001.pdf